CLINICAL TRIAL: NCT07257822
Title: The Digital Diabetes Patient Reminder (DIPAR) Tool to Improve Clinical Outcomes and Process of Management in Adults With Type 2 Diabetes: A Proof-of-Concept Randomized Controlled Trial
Brief Title: The Digital Diabetes Patient Reminder (DIPAR) Tool For Adults With Type 2 Diabetes
Acronym: DIPAR RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: Regionaal Ziekenhuis Heilig Hart Tienen (Other); Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Goderis Geert, Prof. Dr., MD, PhD, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: S70410
Record Dates: First submitted 2025-09-24; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
Keywords: Diabetes; Type 2 Diabetes Mellitus; Self-Care; Self-Management; Digital Intervention; Mobile Health Application; Joint action on cardiovascular diseases and diabetes; JACARDI; The Digital Diabetes Patient Reminder project; DIPAR
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Randomization will be carried out by an external person to the study and the data will be analyzed by an external extension
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DIPAR Intervention Group (Experimental): Standard of Care and the Digital DIPAR Intervention (reminder function + consultation dashboard)
  Interventions: Device: Digital Diabetes Patient Reminder Tool; Other: Standard of Care treatment and follow-up
- Control Group (Other): Standard of Care
  Interventions: Other: Standard of Care treatment and follow-up

INTERVENTIONS:
Device: Digital Diabetes Patient Reminder Tool — - Reminder function: participants will receive reminders that align with the minimal follow-up requirements in Belgium, when the HbA1c and albuminuria measurements are overdue
  o Notification schedule: HbA1c: First reminder after 7 months without a measurement; second reminder 4 weeks later if still overdue.
  Albuminuria: First reminder after 13 months without a measurement; second reminder 4 weeks later if still overdue.
  - Consultation dashboard: this feature will allow the display selected diabetes clinical parameters in a visual and colorful display. The selected parameters are: HbA1c (%), LDL-C (mg/dl), systolic and diastolic blood pressure (mmHg), albuminuria (mg/gACR), eGFR (ml/min/1.73m2) and BMI (weight/lenght2). Furthermore, participants will be provided with a questionnaire that targets selfcare behaviors and are required to complete this before consultations with their diabetes-specialist or general practitioner.
  Arms: DIPAR Intervention Group
Other: Standard of Care treatment and follow-up — This allows for the control to group to receive only their routine consultation and follow-up care as provided by their diabetes specialist.

SUMMARY:
Digital health tools may present an opportunity to address these challenges by enhancing care delivery, improving patient engagement, and facilitating better disease management for chronic diseases such as type 2 diabetes mellitus (T2DM). This primary objective of this randomized controlled trial is to evaluate whether the Diabetes Digital Patient Reminder (DIPAR), embedded in patient portal, can increase the proportion of T2DM patients who have their albuminuria measured at least once annually by either a general practitioner (GP) or a diabetes specialist, as documented in their hospital medical records (EMD), thereby reflecting active monitoring of diabetes-related parameters.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effectiveness of the DIPAR digital tool in improving the management process of patients with type 2 diabetes mellitus (T2DM).

The DIPAR tool consists of two core functionalities designed to support diabetes management: a reminder function and a consultation dashboard.

1. Reminder Function The reminder feature aims to encourage timely diabetes-related clinical follow-ups. It provides patients with automated notifications through the MyNexuzhealth patient portal, usually installed in the mobile phones of the patients, when their measurements for HbA1c and Albuminuria are overdue. These reminders align with the minimal follow-up requirements in Belgium, where HbA1c must be measured biannually and albuminuria annually. We hypothesize that these reminders will prompt patients to schedule routine clinical follow-ups with their general practitioner or diabetes specialist.

   Notification schedule
   * HbA1c: First reminder after 7 months without a measurement; second reminder 4 weeks later if still overdue.
   * Albuminuria: First reminder after 13 months without a measurement; second reminder 4 weeks later if still overdue.
2. Consultation Dashboard

   The consultation dashboard will be provided study participants at the participating institution and will display the following relevant clinical data, extracted from the medical dossier of the diabetes specialist in a visual and colourful display of the progress over time:
   * Clinical outcomes: HbA1c (%), LDL-C (mg/dl), systolic and diastolic blood pressure (mmHg), albuminuria (mg/gACR), eGFR (ml/min/1.73m2) and BMI (weight/lenght2)

   Additionally, the tool includes a questionnaire that patients can complete before consultations to provide insights into their behavior and attitudes toward self-management during the consultations with their physicians. This will include lifestyle-related questions including: medication intake, smoking, weight, fruit and vegetable intake in weekly diet, intake of sugary snacks and drinks, weekly physical activity, and whether or not diabetic foot and fundoscopy examination have occurred.

   The trial will be conducted in two phases. In Phase 1, participants in the intervention group will have access to the reminder function of the DIPAR extension. In Phase 2, they will additionally use the consultation dashboard alongside their diabetes specialist, while retaining access to the reminder function. This phased approach ensures a gradual introduction of the tool, reduces complexity for participants, and allows assessment of the reminder function's impact on diabetes management processes before incorporating the dashboard.

   Research Question Does the use of the DIPAR tool improve the measurement and documentation of clinical parameters and increase adherence to recommended diabetes care, particularly the measurement of albuminuria in individuals with T2DM?

   Primary Objective The primary objective is to assess whether the implementation of the DIPAR tool can increase the proportion of patients who receive at least one annual measurement of albuminuria, performed either by the general practitioner (GP) or a diabetes specialist, as documented in the electronic medical record (EMD), thereby reflecting improved monitoring of diabetes-related parameters.

   Secondary Objectives The key secondary objective is to assess whether the proportion of patients with at least two documented HbA1c measurements in the EMD reports of the GP or diabetes specialist increases with the use of the DIPAR tool.

   The exploratory secondary objectives are:

   • To determine the proportion of patients with T2DM who have their HbA1c measurements documented in the EMD of i. the general practitioner and ii. the diabetes specialist.
   * To explore the perceived usability and acceptability of the digital tool among both patients and healthcare providers, as well as its potential to improve health literacy in patients within the intervention group.
   * To evaluate changes in key diabetes-related clinical parameters, specifically HbA1c, albuminuria, LDL-cholesterol, and blood pressure over the study duration.

   Study Duration

   The study is expected to last approximately 15 months (October 2025-January 2027). Key activities are planned as follows:
   * October-December 2025

     * Site preparations at both centers.
     * Participant recruitment, informed consent collection, baseline questionnaires, and randomization.
   * December 2025-December 2026

     o Intervention phase (12 months per participant, starting immediately after randomization).

     o Intervention group receives access to the DIPAR reminder function.

     o Clinical follow-up visits at 6 and 12 months serve as primary data collection points.

     o Six months after study start, intervention group gains access to the DIPAR consultation dashboard for use during physician visits.
   * Final 3 months of intervention (October-December 2026)

     o Invitation of participants from the intervention group to semi-structured interviews or focus groups with healthcare providers.

     o Completion of the Dutch version of the mHealth App Usability Questionnaire (MAUQ), submitted electronically or on paper.
   * January 2027 Final data collection and study close-out.

   Each participant will be involved for approximately 12 months; for those invited to the qualitative assessments, participation may extend to 14-15 months.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent of the participant or their legally authorized representative has been obtained prior to any screening procedures;
* Adults 18 years or older;
* Treated and followed-up for Type 2 diabetes at the department of endocrinology at the participating hospitals;
* Patients with (the ability to access) the MyNexuz patient portal;
* Patients with the ability to understand Dutch, French or English.

Exclusion Criteria:

* Participant is pregnant or hospitalized at the time of recruitment;
* Are unable to use a mobile phone because of mental or cognitive impairment;
* Deemed ineligible by the treating physicians.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Documentation rate of Albuminuria | 12 months post intervention
  Defining the proportion of patients with at least one measured and documented albuminuria value in the electronic medical dossier

SECONDARY OUTCOMES:
Documentation rate of HbA1c (2x) | 12 month post intervention
  Defining the proportion of patients with at least two measured and documented HbA1c value in the electronic medical dossier
Documentation rate of HbA1c (1x) | 12 month post intervention
  Defining the proportion of patients with at least one measured and documented HbA1c value in the electronic medical dossier
DIPAR Usability | 12 months post intervention
  With the validated mHealth App Usability Questionnaire the usability of DIPAR will be assessed.
  Scale Title: mHealth App Usability Questionnaire (21 items) Response scale: With 5-point Likert scale
  1 = strongly disagree, 5=strongly agree and 0=Not Applicable
DIPAR Acceptability | 12 months post intervention
  Semi structured interviews and focus group discussions are two qualitative research methodology that will be employed to assess the acceptability of the DIPAR tool by patients and physicians
Change in HbA1c | Baseline, Month 6 and Month 12 post intervention
  * Change of these clinical parameters after 6 months from baseline
  * Change of these clinical parameters after 12 months from baseline
Change in Albuminuria | Baseline, Month 6 and Month 12 post intervention
  * Change of these clinical parameters after 6 months from baseline
  * Change of these clinical parameters after 12 months from baseline
Change in Cholesterol | Baseline, Month 6 and Month 12 post intervention
  * Change of these clinical parameters after 6 months from baseline
  * Change of these clinical parameters after 12 months from baseline
Change in Blood Pressure | Baseline, Month 6 and Month 12 post intervention
  * Change of these clinical parameters after 6 months from baseline
  * Change of these clinical parameters after 12 months from baseline
Change in Weight | Baseline, Month 6 and Month 12 post intervention
  * Change of these clinical parameters after 6 months from baseline
  * Change of these clinical parameters after 12 months from baseline
Change in Heart rate | Baseline, Month 6 and Month 12 post intervention
  * Change of these clinical parameters after 6 months from baseline
  * Change of these clinical parameters after 12 months from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Roman Vangoitsenhoven, Prof Dr., Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (2):
- Belgium (2):
  - Regional Hospital of Leuven, Leuven, Flemish Brabant
  - University Hospital of UZ Leuven, Leuven, Flemish Brabant

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: This is the official website for the trial and DIPAR project — https://gbiomed.kuleuven.be/english/research/50000687/50000695/NL/jacardi-eng/home